CLINICAL TRIAL: NCT04779476
Title: Effectiveness of Alveogyl and Cutanplast Dressing on Postoperative Pain Following Tooth Extraction: A Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Ahmad Assari, Dr. Ahmad Assari, Riyadh Elm University
Other Study IDs: FRP/2021/319
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Facial Pain; Pain, Postoperative; Pain, Orofacial
Keywords: Alveogyl; Eugenol; Dental extraction; Post extraction pain
MeSH Terms: conditions — Facial Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: No dressing material will be used post dental extraction
- Alveogyl Group: Alveogyl will be placed in the dental socket after extraction
  Interventions: Other: Socket Dressing
- Cutanplast Group: Absorbable gelatin sponges contain will be placed in the dental socket after extraction
  Interventions: Other: Socket Dressing

INTERVENTIONS:
Other: Socket Dressing — Following dental extraction immediately, the socket will be dressed with one of the materials tested
  Groups: Alveogyl Group; Cutanplast Group

SUMMARY:
This study aims to assess the post-dental extraction pain following the application of two different dressing materials.

Alvogyl® and Absorbable gelatin sponges

DETAILED DESCRIPTION:
Effective postoperative pain relief improves the quality of recovery and the resumption of normal activities. Many options are available for postoperative pain relief following tooth extraction including systemic analgesic, intra-alveolar socket dressing medicaments, and follow the postoperative instructions; the choice of the medication determined by drug availability, chance of side effect of some drugs and financial considerations. The use of intra-alveolar dressing materials is widely suggested in the literature such as Alvogyl® that used as palliative treatment which includes eugenol (analgesic, anti-inflammatory), iodoform (antimicrobial), and butamen (anesthetic). Absorbable gelatin sponges contain haemostatic material and may be used for local application in surgical procedures where traditional haemostasis is difficult. In addition to its haemostatic effect, an absorbable gelatin sponge can be used as a drug reservoir to provide sustained release of drugs

The aim of this study is to measure the pain intensity after using socket dressing materials following tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Single tooth extraction
* Upper and lower teeth

Exclusion Criteria:

* Surgical extraction
* Medically compromised patients
* Presence of active infection
* Presence of pathology

Ages: 13 Years to 22 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients referred from the orthodontic department for extraction of p
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
3 hrs post extraction pain | three hours after the extraction
  Visual analogue scale score for pain
6 hrs post extraction pain | six hours after the extraction
  Visual analogue scale score for pain
12 hrs post extraction pain | twelve hours after the extraction
  Visual analogue scale score for pain
24 hrs post extraction pain | twenty-four hours after the extraction
  Visual analogue scale score for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Assari, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The anticipated number may not be reached

REFERENCES:
- [Result] Bloomer CR. Alveolar osteitis prevention by immediate placement of medicated packing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Sep;90(3):282-4. doi: 10.1067/moe.2000.108919. PMID 10982947
- [Result] Summers L, Matz LR. Extraction wound sockets. Histological changes and paste packs--a trial. Br Dent J. 1976 Dec 21;141(12):377-9. doi: 10.1038/sj.bdj.4803851. No abstract available. PMID 1070322
- [Result] Kaur G, Athar M, Alam MS. Eugenol precludes cutaneous chemical carcinogenesis in mouse by preventing oxidative stress and inflammation and by inducing apoptosis. Mol Carcinog. 2010 Mar;49(3):290-301. doi: 10.1002/mc.20601. PMID 20043298
- [Result] Kafali H, Iltemur Duvan C, Gozdemir E, Simavli S, Ozturk Turhan N. Placement of bupivacaine-soaked Spongostan in episiotomy bed is effective treatment modality for episiotomy-associated pain. J Minim Invasive Gynecol. 2008 Nov-Dec;15(6):719-22. doi: 10.1016/j.jmig.2008.08.006. PMID 18971135